CLINICAL TRIAL: NCT03707379
Title: The Effect of Share Care Model in the Improvement of Diabetes Management
Status: Recruiting | Type: Observational
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 【2016】004
Record Dates: First submitted 2018-07-23; First posted 2018-10-16 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes mellitus; Diabetic management; Share care
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- common care group: diabetic patients under common care group

SUMMARY:
The situation of diabetes management in China is serious. To set up hierarchical medical system is necessary, though there was no mature or effective diabetes management model in the mainland. To explore a new path for hierarchical medical system, we would localize the share care model of diabetes management in Taiwan. Diabetic experts, diabetic educators and community doctors would use interactive information platform and self-glucose monitor with application on mobile phone to manage diabetic patients together. The model will be applied in six diabetic centers, and patients we will be managed in the new model and followed, and at the same time patients that managed in the conventional model in the real world, the differences of proportion who achieve a composite goal will be compared yearly for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients

Exclusion Criteria:

* Patients had not signed the consent form
* Patients with sever hart failure, hepatic failure, renal failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients in Ruijing Diabetes Hospital
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2016-03-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 1 year
  control rate of HbA1c<7.0%

SECONDARY OUTCOMES:
blood pressure | 1 year
  control rate of blood pressure<140/90 millimetres of mercury
LDL-C | 1 year
  control rate of LDL-C<2.6mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhong Xiao, Study Director — Beijing Tsinghua Changgeng Hospital
Locations (1):
- Beijing Ruijing Diabetes Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] An L, Wang Y, Cao C, Chen T, Zhang Y, Chen L, Ren S, Tang M, Ma F, Li X, Yuan S, Zhao W, Lee Y, Xiao J. Screening cardiovascular risk factors of diabetes patients in the primary diabetes clinics. Medicine (Baltimore). 2021 Jul 30;100(30):e26722. doi: 10.1097/MD.0000000000026722. PMID 34397707